CLINICAL TRIAL: NCT03544034
Title: Partnering With Patients for Improving Medication Safety During Transitions of Care: Implications for Work System Design
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Johns Hopkins University (Other)
Collaborators: The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00175392
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Patient Safety; Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: A pre-post study in two hospitals. Implementation will be done at the organization level (for all 65 and older patients admitted to hospitalist service in these two hospitals.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Routine/ standard care and retrospective chart review for identifying preventable and ameliorable Adverse drug events as baseline
- Post-intervention (Experimental): Hometeam toolkit interventions (including improved discharge education, proactive medication safety assessment in daily rounds and handoffs, safety briefings) applied in all hospitalist services.
  Interventions: Behavioral: HomeTeam Toolkit

INTERVENTIONS:
Behavioral: HomeTeam Toolkit — A multi-component intervention (8S's)
  1. Safety at home through partnership.
  2. Safety risk assessment at the admission
  3. Safety agenda setting for coordinating efforts among professionals to prepare patient/ family for self-management
  4. Safety tools. Cognitive tools to support patient/family after discharge
  5. Safety education. Enhanced Patient/ family medication safety education
  6. Safety briefings with patient/family A mechanism to proactively address common and patient/family specific risks.
  7. Safety through learning routines across the care continuum
  8. Safety assessment after discharge
  Arms: Post-intervention

SUMMARY:
This project is to develop, implement, pilot evaluate, and disseminate a medication safety program (HomeTeam) that consolidates strategies to help patients by partnering with patients and their informal caregivers during transitions from hospital to home. Care transitions, especially from hospital to home, are high-risk periods for medication errors, and are frequently associated with serious adverse drug events (ADEs) and preventable readmissions. Older adults with multi-morbid conditions who have complex medication regimes are especially prone to these risks. Patients and family caregivers may experience a dramatic transition in roles and responsibilities immediately after hospital discharge. Patients and family caregivers are relatively passive recipients in their care and medication management in the hospital, but when patients arrive at home, patients have the primary responsibility for their care and medication use (with professional care providers switching to a 'supporting' function). Although this significant transition in the nature and intensity of patient work needs to be managed actively, often patients and family members are not adequately engaged and prepared in the hospital, and not effectively supported for safe medication use after hospital discharge. More specifically, patients and family members may not understand essential steps in the management of their condition, and have difficulty contacting appropriate health care practitioners for guidance. Although most organizations deploy multiple layers of interventions for improving care transitions, reducing postdischarge adverse drug events (ADEs), 30-day readmissions and emergency department (ED) visits, their impact to date has been small, and there remains significant and urgent need to fundamentally redesign the hospital-to-home care transition process. Investigators believe that one practical and potentially effective way for this 'much-needed' redesign is through engaging and supporting patients and families in safe medication use. Investigators' proposed program 'HomeTeam' will contain evidence-based tools and methods for engaging patients and shifting culture towards a truly patient-centered care for medication safety.

DETAILED DESCRIPTION:
The 'HomeTeam will be developed and evaluated by completing 3 specific aims:

Aim #1: Develop components of a multi-faceted program (HomeTeam) that consolidates evidence-based practices in patient and family activation and engagement related to medication safety, with the goal to adequately and reliably support transitions from the hospital to the patient home "work system" for medication management. Inpatient stays and the hospital discharge periods will be targeted as opportunities in activating, engaging, and enabling patients and family members to improve medication safety.

(1a) Identify evidence-based practices in patient and family activation and engagement related to medication safety during care transitions.

1. b) Develop program components (e.g., action-oriented patient/ family education, improved medication reconciliation, patient-centered rounds, learning systems through systematic feedback from home care professionals)-including tools to assess, prioritize, streamline, and integrate existing practices- aimed at engaging patients and families and supporting medication use safety during care transitions from hospital to home with a participatory design (PD) approach.

   Aim #2: Refine and implement the HomeTeam program in two organizations (one academic, one community hospital), with a peer-to-peer assessment methodology to identify and refine patient and family engagement practices for transitional care medication safety.
2. a) Refine HomeTeam program through participatory design approach and peer-to-peer assessment

(2b) Implement and pilot test HomeTeam in all participating sites

Aim #3: Evaluate the implementation process and the impact of the toolkit 'HomeTeam' on medication safety after hospital discharge. Investigators will use a pre-post design to evaluate the impact of the toolkit over a one year period, focusing on 65 years of age and older medicine patients. The primary outcome is preventable and ameliorable adverse drug events (ADEs) after discharge. Secondary outcomes include 30-day post-discharge readmissions and ED visits due to medication-related issues process improvement assessment, patient-reported outcomes, and toolkit adoption assessment (e.g., acceptability, feasibility). Qualitative methods (post-implementation interviews with clinicians and patient/ family members) will be used as part of the evaluation.

Hypothesis: Investigators hypothesize that the HomeTeam Medication Safety Program will reduce preventable and ameliorable post-discharge 30-day ADEs in the following subpopulations: older adults with at least 5 medications discharged from hospital to home on (H01) anticoagulants, (H0b) opioids, (H0c) diabetes agents.

The project will be conducted in two hospitals: Bayview Medical Center (academic) and Howard County Medical Center (community). Dissemination plans include national medication safety organizations (e.g., Institute for Safe Medication Practices), patient safety organizations (e.g., Batz Patient Safety Foundation), and professional societies (e.g., Society of Hospital Medicine). Different dissemination modalities are planned, including story-telling through social media and short videos targeted for patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* medicine patients
* hospitalized from home
* English speaking
* no cognitive problems/ can consent

Exclusion Criteria:

* surgery patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Preventable adverse drug events | 30 days after hospital discharge
  Preventable ADEs are injuries that could have bee n avoided, that is, an injury judged to probably be the result of an error or a system design flaw.
Ameliorable adverse drug events | 30 days after hospital discharge
  Ameliorable ADEs are injuries whose severity could have been substantially reduced if different actions or procedures had been performed or followed.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Gurses, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Univ Armstrong Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No